CLINICAL TRIAL: NCT00784043
Title: Longitudinal Efficacy in Young Children Implanted Bilaterally With MED-EL COMBI 40+ / PULSARCI100/SONATATI100 Cochlear Implant Systems.
Brief Title: Bilateral Cochlear Implantation in Children With the MED-EL Cochlear Implant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-EL NA 013
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Hearing Loss
Keywords: Cochlear implant; hearing loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral (Experimental): Bilaterally implanted simultaneously
  Interventions: Device: Cochlear Implant
- Unilateral (Experimental): Unilaterally implanted
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — Bilateral Implantation in children
  Other Names: MED-EL Cochlear Implant; Combi 40+; PulsarCI100; SonataTI100

SUMMARY:
The purpose of this study is to evaluate and document longitudinal efficacy in young children implanted bilaterally with MED-EL COMBI 40+ / PULSARCI100/SONATATI100 cochlear implant systems.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 36 months of age at time of implantation
* Profound bilateral sensorineural hearing loss
* English as the primary language in the home
* Realistic expectations of guardians
* Child must be enrolled in a post-operative rehabilitative/educational program that supports the use of cochlear implants and the development of auditory-based skills
* Willing and available to comply with all scheduled procedures as defined in the protocol

Audiological:

* Profound bilateral sensorineural hearing loss with average thresholds between ears of 90 dB HL or greater at 1000 Hz and above, and must demonstrate minimal functional benefit from conventional amplification
* Behavioral test measures must include unaided threshold measures for the right and left ears using insert earphones; left-alone and right-alone aided sound field threshold measurements; and aided and unaided speech-awareness / detection thresholds (for each ear individually)
* Children accepted into the study must be able to demonstrate a consistent response to sound. If a child has no measurable hearing, he/she must be able to demonstrate a consistent response to vibrotactile stimuli.
* All children must have completed an appropriate trial period with optimally fit amplification prior to inclusion in the study.

Medical:

* Good general health status, as judged by Primary Investigator
* Patent cochleae bilaterally, as indicated by radiological evaluation
* No contraindications for surgery, in general, or cochlear implant surgery in particular

Exclusion Criteria:

* Prior experience with any cochlear implant system
* Younger than 12 months or older than 36 months at time of implantation
* Audiological: Presence of otoacoustic emissions and/or cochlear microphonic, indicating possible condition of auditory neuropathy

Medical:

* Evidence of ossification that would prevent full insertion of the standard C40+ / PULSARCI100 /SONATATI100 electrode array in the cochlea(e) to be implanted, as indicated by radiological evaluation
* Abnormal or malformed cochlea(e) to be implanted
* Severed or non-functional auditory nerve in the ear(s) to be implanted
* Central auditory lesion
* Cognitive and/or neurological dysfunction
* Auditory neuropathy

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2004-03; Primary Completion 2009-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dallas Otolaryngology Associates, Dallas, Texas
  - Callier Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Kuhn-Inacker H, Shehata-Dieler W, Muller J, Helms J. Bilateral cochlear implants: a way to optimize auditory perception abilities in deaf children? Int J Pediatr Otorhinolaryngol. 2004 Oct;68(10):1257-66. doi: 10.1016/j.ijporl.2004.04.029. PMID 15364496
- [Background] Nopp P, Schleich P, D'Haese P. Sound localization in bilateral users of MED-EL COMBI 40/40+ cochlear implants. Ear Hear. 2004 Jun;25(3):205-14. doi: 10.1097/01.aud.0000130793.20444.50. PMID 15179112
- [Background] Schleich P, Nopp P, D'Haese P. Head shadow, squelch, and summation effects in bilateral users of the MED-EL COMBI 40/40+ cochlear implant. Ear Hear. 2004 Jun;25(3):197-204. doi: 10.1097/01.aud.0000130792.43315.97. PMID 15179111
- [Background] Muller J, Schon F, Helms J. Speech understanding in quiet and noise in bilateral users of the MED-EL COMBI 40/40+ cochlear implant system. Ear Hear. 2002 Jun;23(3):198-206. doi: 10.1097/00003446-200206000-00004. PMID 12072612
- [Background] Schon F, Muller J, Helms J. Speech reception thresholds obtained in a symmetrical four-loudspeaker arrangement from bilateral users of MED-EL cochlear implants. Otol Neurotol. 2002 Sep;23(5):710-4. doi: 10.1097/00129492-200209000-00018. PMID 12218624
- [Background] Tyler RS, Gantz BJ, Rubinstein JT, Wilson BS, Parkinson AJ, Wolaver A, Preece JP, Witt S, Lowder MW. Three-month results with bilateral cochlear implants. Ear Hear. 2002 Feb;23(1 Suppl):80S-89S. doi: 10.1097/00003446-200202001-00010. PMID 11883771
- [Background] Winkler F, Schon F, Peklo L, Muller J, Feinen Ch, Helms J. [The Wurzburg questionnaire for assessing the quality of hearing in CI-children (WH-CIK)]. Laryngorhinootologie. 2002 Mar;81(3):211-6. doi: 10.1055/s-2002-25042. German. PMID 11967774
- [Background] Zimmerman-Phillips S, Robbins AM, Osberger MJ. Assessing cochlear implant benefit in very young children. Ann Otol Rhinol Laryngol Suppl. 2000 Dec;185:42-3. doi: 10.1177/0003489400109s1217. No abstract available. PMID 11140998
- [Background] Kirk KI, Pisoni DB, Osberger MJ. Lexical effects on spoken word recognition by pediatric cochlear implant users. Ear Hear. 1995 Oct;16(5):470-81. doi: 10.1097/00003446-199510000-00004. PMID 8654902
- [Background] Grantham DW, Ashmead DH, Ricketts TA, Labadie RF, Haynes DS. Horizontal-plane localization of noise and speech signals by postlingually deafened adults fitted with bilateral cochlear implants. Ear Hear. 2007 Aug;28(4):524-41. doi: 10.1097/AUD.0b013e31806dc21a. PMID 17609614
- [Background] Ricketts TA, Grantham DW, Ashmead DH, Haynes DS, Labadie RF. Speech recognition for unilateral and bilateral cochlear implant modes in the presence of uncorrelated noise sources. Ear Hear. 2006 Dec;27(6):763-73. doi: 10.1097/01.aud.0000240814.27151.b9. PMID 17086085
- [Background] Dorman MF, Dahlstrom L. Speech understanding by cochlear-implant patients with different left- and right-ear electrode arrays. Ear Hear. 2004 Apr;25(2):191-4. doi: 10.1097/01.aud.0000120367.70123.9a. PMID 15064664
- [Background] Laback B, Pok SM, Baumgartner WD, Deutsch WA, Schmid K. Sensitivity to interaural level and envelope time differences of two bilateral cochlear implant listeners using clinical sound processors. Ear Hear. 2004 Oct;25(5):488-500. doi: 10.1097/01.aud.0000145124.85517.e8. PMID 15599195
- [Background] Van Hoesel R, Ramsden R, Odriscoll M. Sound-direction identification, interaural time delay discrimination, and speech intelligibility advantages in noise for a bilateral cochlear implant user. Ear Hear. 2002 Apr;23(2):137-49. doi: 10.1097/00003446-200204000-00006. PMID 11951849
- [Background] Pijl S. Single-channel versus bilateral multichannel cochlear implant results: a case report. Ear Hear. 1991 Dec;12(6):431-3. doi: 10.1097/00003446-199112000-00007. PMID 1797610
- [Background] Beijen JW, Snik AF, Mylanus EA. Sound localization ability of young children with bilateral cochlear implants. Otol Neurotol. 2007 Jun;28(4):479-85. doi: 10.1097/MAO.0b013e3180430179. PMID 17473710
- [Background] Truy E, Ionescu E, Ceruse P, Gallego S. The binaural digisonic cochlear implant: surgical technique. Otol Neurotol. 2002 Sep;23(5):704-9. doi: 10.1097/00129492-200209000-00017. PMID 12218623
- [Background] Brown KD, Balkany TJ. Benefits of bilateral cochlear implantation: a review. Curr Opin Otolaryngol Head Neck Surg. 2007 Oct;15(5):315-8. doi: 10.1097/MOO.0b013e3282ef3d3e. PMID 17823546
- [Background] Das S, Buchman CA. Bilateral cochlear implantation: current concepts. Curr Opin Otolaryngol Head Neck Surg. 2005 Oct;13(5):290-3. doi: 10.1097/01.moo.0000179808.00638.ab. PMID 16160523
- [Background] Offeciers E, Morera C, Muller J, Huarte A, Shallop J, Cavalle L. International consensus on bilateral cochlear implants and bimodal stimulation. Acta Otolaryngol. 2005 Sep;125(9):918-9. doi: 10.1080/00016480510044412. No abstract available. PMID 16109670
- [Background] Verschuur CA, Lutman ME, Ramsden R, Greenham P, O'Driscoll M. Auditory localization abilities in bilateral cochlear implant recipients. Otol Neurotol. 2005 Sep;26(5):965-71. doi: 10.1097/01.mao.0000185073.81070.07. PMID 16151344
- [Background] Senn P, Kompis M, Vischer M, Haeusler R. Minimum audible angle, just noticeable interaural differences and speech intelligibility with bilateral cochlear implants using clinical speech processors. Audiol Neurootol. 2005 Nov-Dec;10(6):342-52. doi: 10.1159/000087351. Epub 2005 Aug 5. PMID 16103645
- [Background] Sharma A, Dorman MF, Kral A. The influence of a sensitive period on central auditory development in children with unilateral and bilateral cochlear implants. Hear Res. 2005 May;203(1-2):134-43. doi: 10.1016/j.heares.2004.12.010. PMID 15855038
- [Background] Laszig R, Aschendorff A, Stecker M, Muller-Deile J, Maune S, Dillier N, Weber B, Hey M, Begall K, Lenarz T, Battmer RD, Bohm M, Steffens T, Strutz J, Linder T, Probst R, Allum J, Westhofen M, Doering W. Benefits of bilateral electrical stimulation with the nucleus cochlear implant in adults: 6-month postoperative results. Otol Neurotol. 2004 Nov;25(6):958-68. doi: 10.1097/00129492-200411000-00016. PMID 15547426
- [Background] Litovsky RY, Parkinson A, Arcaroli J, Peters R, Lake J, Johnstone P, Yu G. Bilateral cochlear implants in adults and children. Arch Otolaryngol Head Neck Surg. 2004 May;130(5):648-55. doi: 10.1001/archotol.130.5.648. PMID 15148192
- [Background] Schauwers K, Gillis S, Daemers K, De Beukelaer C, De Ceulaer G, Yperman M, Govaerts PJ. Normal hearing and language development in a deaf-born child. Otol Neurotol. 2004 Nov;25(6):924-9. doi: 10.1097/00129492-200411000-00011. PMID 15547421
- [Background] Seeber BU, Baumann U, Fastl H. Localization ability with bimodal hearing aids and bilateral cochlear implants. J Acoust Soc Am. 2004 Sep;116(3):1698-709. doi: 10.1121/1.1776192. PMID 15478437
- [Background] Stark T, Engel A, Borkowski G. [Bilateral cochlea implantation in varying duration of deafness]. Laryngorhinootologie. 2004 Jan;83(1):20-2. doi: 10.1055/s-2004-814097. German. PMID 14740301
- [Background] Tyler RS, Witt SA, Dunn CC. Trade-offs between better hearing and better cosmetics. Am J Audiol. 2004 Dec;13(2):193-9. doi: 10.1044/1059-0889(2004/024). PMID 15903145
- [Background] van Hoesel RJ. Exploring the benefits of bilateral cochlear implants. Audiol Neurootol. 2004 Jul-Aug;9(4):234-46. doi: 10.1159/000078393. PMID 15205551
- [Background] Au DK, Hui Y, Wei WI. Superiority of bilateral cochlear implantation over unilateral cochlear implantation in tone discrimination in chinese patients. Am J Otolaryngol. 2003 Jan-Feb;24(1):19-23. doi: 10.1053/ajot.2003.8. PMID 12579478
- [Background] Kong W, Yu L, Xu Y, Yue J, Xiong X, Zhu L, Duan J. [Benefit of bilateral cochlear implantation on congenital prelingually deafened Chinese-speaking children]. Lin Chuang Er Bi Yan Hou Ke Za Zhi. 2003 Oct;17(10):577-9. Chinese. PMID 14727421
- [Background] Caleffe-Schenck, N, Franz, D. (2004). Checklist of Auditory Communication Skills. Volta Review 104(3): 175-196.
- [Background] Semel, E, Wiig, E, Secord, W. (2003). Clinical Evaluation of Language Fundamentals Fourth Edition. San Antonio, Texas: The Psychological Corporation
- [Background] Stark, T, Müller, J, Vischer, M, Schön, F, Senn, P, Engel, A, Kompis, M, Hildmann, H, Helms, J. (2002). Multicenter study on bilateral cochlear implantation. In Kubo, T, Takahashi, Y, Iwaki, T, (eds.) Cochlear implants - an update. The Hague: Kugler.
- [Background] Goldman, R, Fristoe, M. (2000). Goldman-Fristoe Test of Articulation Second Edition. Circle Pines, Minnesota: American Guidance Service.
- [Background] In Kim, C, Chang, S, Lim, D, (eds). Updates in cochlear implantation. Adv. Otorhinolarygol, Basel: Karger.
- [Background] Lawson, D, Wilson, B, Zerbi, M, Finley, C. (1999). Fourth quarterly progress report: Speech processors for auditory prostheses. NIH Contract N01-DC-8-2105.
- [Background] Schön, F, Mueller, J, Helms, J. (1999). Results of bilateral cochlear implantation. European Archives of Oto-Rhino-Laryngology 156:106.
- [Background] Lawson, D, Zerbi, M, Wilson, B. (1998). First quarterly progress report: Speech processors for auditory prostheses. NIH Contract N01-DC-8-2105.
- [Background] Dunn, L, Dunn, L. (1997). Peabody Picture Vocabulary Test Third Edition. Circle Pines, Minnesota: American Guidance Service.
- [Background] Williams, K. (1997). Expressive Vocabulary Test. Circle Pines, Minnesota: American Guidance Service.
- [Background] Kaufman, N. (1995). Kaufman Speech Praxis Test for Children. Detroit, Michigan: Wayne State University Press.
- [Background] Fenson, L, Dale, P, Resnick, J, Thal, D, Bates, E, Hartung, J, Pethick, S, Reilly, J. (1993). MacArthur Communicative Development Inventories: User's Guide and Technical Manual. Baltimore, Maryland: Paul H. Brokes Publishing Company.
- [Background] Reynell, J, Gruber, C. (1990). Reynell Developmental Language Scales. Los Angeles, California: Western Psychological Services.
- [Background] Jerger, S, Jerger, J. (1984). Pediatric Speech Intelligibility Test. St. Louis, Missouri: Auditec of St. Louis.
- [Background] Erber, N. (1982). Auditory Training. Washington, DC: Alexander Graham Bell Association.
- [Background] Haskins, H. (1949). A phonetically balanced test of speech discrimination for children. Master's Theis. Northwestern University, Evanston, Illinois.
- [Background] Ramsden R, Greenham P, O'Driscoll M, Mawman D, Proops D, Craddock L, Fielden C, Graham J, Meerton L, Verschuur C, Toner J, McAnallen C, Osborne J, Doran M, Gray R, Pickerill M. Evaluation of bilaterally implanted adult subjects with the nucleus 24 cochlear implant system. Otol Neurotol. 2005 Sep;26(5):988-98. doi: 10.1097/01.mao.0000185075.58199.22. PMID 16151348
- [Background] Schoen F, Mueller J, Helms J, Nopp P. Sound localization and sensitivity to interaural cues in bilateral users of the Med-El Combi 40/40+cochlear implant system. Otol Neurotol. 2005 May;26(3):429-37. doi: 10.1097/01.mao.0000169772.16045.86. PMID 15891645
- [Background] Long CJ, Eddington DK, Colburn HS, Rabinowitz WM. Binaural sensitivity as a function of interaural electrode position with a bilateral cochlear implant user. J Acoust Soc Am. 2003 Sep;114(3):1565-74. doi: 10.1121/1.1603765. PMID 14514210
- [Background] Tyler RS, Dunn CC, Witt SA, Preece JP. Update on bilateral cochlear implantation. Curr Opin Otolaryngol Head Neck Surg. 2003 Oct;11(5):388-93. doi: 10.1097/00020840-200310000-00014. PMID 14502072
- [Background] van Hoesel RJ, Tyler RS. Speech perception, localization, and lateralization with bilateral cochlear implants. J Acoust Soc Am. 2003 Mar;113(3):1617-30. doi: 10.1121/1.1539520. PMID 12656396
- [Background] Vermeire K, Brokx JP, Van de Heyning PH, Cochet E, Carpentier H. Bilateral cochlear implantation in children. Int J Pediatr Otorhinolaryngol. 2003 Jan;67(1):67-70. doi: 10.1016/s0165-5876(02)00286-0. PMID 12560152
- [Background] Wilson BS, Lawson DT, Muller JM, Tyler RS, Kiefer J. Cochlear implants: some likely next steps. Annu Rev Biomed Eng. 2003;5:207-49. doi: 10.1146/annurev.bioeng.5.040202.121645. Epub 2003 Apr 16. PMID 12704085
- [Background] Au, D., Hui, Y., Wei, W, & Wong, B. (2002). Speech recognition between bilaterally and unilaterally cochlear implanted and hearing aid fitted users. In Kubo, T., Takahashi Y., & Iwaki, T. (Ed.) Cochlear implants - an update. The Hague: Kugler.
- [Background] Gantz BJ, Tyler RS, Rubinstein JT, Wolaver A, Lowder M, Abbas P, Brown C, Hughes M, Preece JP. Binaural cochlear implants placed during the same operation. Otol Neurotol. 2002 Mar;23(2):169-80. doi: 10.1097/00129492-200203000-00012. PMID 11875346
- [Background] Summerfield AQ, Marshall DH, Barton GR, Bloor KE. A cost-utility scenario analysis of bilateral cochlear implantation. Arch Otolaryngol Head Neck Surg. 2002 Nov;128(11):1255-62. doi: 10.1001/archotol.128.11.1255. PMID 12431166
- [Background] Mawman DJ, Ramsden RT, O'Driscoll M, Adams T, Saeed SR. Bilateral cochlear implantation--a case report. Adv Otorhinolaryngol. 2000;57:360-3. doi: 10.1159/000059132. No abstract available. PMID 11892189
- [Background] Mueller J, Schoen F, Helms J. Bilateral cochlear implant--new aspects for the future? Adv Otorhinolaryngol. 2000;57:22-7. doi: 10.1159/000059172. No abstract available. PMID 11892152
- [Background] Lawson, D., Wilson, B., Zerbi, M., & Finley, C. (1999). Fourth Quarterly Progress Report. NIH Contract N01-DC-8-2105. Retrieved from http://npp.ninds.nih.gov/ProgressReports/Speech ProcessorsforAuditoryProstheses%20DC82105/SpeechProcessorsWilson4DC82105.pdf
- [Background] van Hoesel, R. J. M., & Clark, G. M. (1999). Speech results with a bilateral multi-channel cochlear implant subject for spatially separated signal and noise. Australian Journal of Audiology, 21, 23-28.
- [Background] Müller, J., Schön, F., & Helms J. (1998). Binaural cochlear implantation: a case report discussing preliminary results. European Archives of Oto-Rhino-Laryngology, 255, 38.
- [Background] Lawson DT, Wilson BS, Zerbi M, van den Honert C, Finley CC, Farmer JC Jr, McElveen JT Jr, Roush PA. Bilateral cochlear implants controlled by a single speech processor. Am J Otol. 1998 Nov;19(6):758-61. PMID 9831150
- [Background] Lawson, D., Zerbi, M., & Wilson, B. (1998). First Quarterly Progress Report. NIH Contract N01-DC-8-2105. Retrieved from http://npp.ninds.nih.gov/ProgressReports/SpeechProcessorsfor AuditoryProstheses%20DC82105/qpr1/qpr1a.html
- [Background] van Hoesel RJ, Clark GM. Psychophysical studies with two binaural cochlear implant subjects. J Acoust Soc Am. 1997 Jul;102(1):495-507. doi: 10.1121/1.419611. PMID 9228813
- [Background] Lawson, D., Wilson, B., Zerbi, M., & Finley, C. (1996). Fifth Quarterly Progress Report. NIH Contract N01-DC-5-2103. Retrieved from http://npp.ninds.nih.gov/ProgressReports/Speech ProcessorsforAuditoryProstheses%20DC52103/qpr5/qpr5.html.
- [Background] Van Hoesel RJ, Clark GM. Fusion and lateralization study with two binaural cochlear implant patients. Ann Otol Rhinol Laryngol Suppl. 1995 Sep;166:233-5. PMID 7668650
- [Background] van Hoesel RJ, Tong YC, Hollow RD, Clark GM. Psychophysical and speech perception studies: a case report on a binaural cochlear implant subject. J Acoust Soc Am. 1993 Dec;94(6):3178-89. doi: 10.1121/1.407223. PMID 8300953
- [Background] Green JD Jr, Mills DM, Bell BA, Luxford WM, Tonokawa LL. Binaural cochlear implants. Am J Otol. 1992 Nov;13(6):502-6. PMID 1449175
- [Background] Pelizzone M, Kasper A, Montandon P. Binaural interaction in a cochlear implant patient. Hear Res. 1990 Oct;48(3):287-90. doi: 10.1016/0378-5955(90)90069-2. PMID 2272938
- [Background] Balkany T, Boggess W, Dinner B. Binaural cochlear implantation: comparison of 3M/House and Nucleus 22 devices with evidence of sensory integration. Laryngoscope. 1988 Oct;98(10):1040-3. doi: 10.1288/00005537-198810000-00002. PMID 3172948

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral | Unilateral
Started | 31 | 6
Completed | 0 | 0
Not Completed | 31 | 6
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Protocol Terminated | 23 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilateral | Unilateral | Total
Number analyzed (Participants) | 31 | 6 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 6 | 37
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information not available for 3 participants.
  Participants
    number analyzed (Participants) | 28 | 6 | 34
    Female | 12 | 0 | 12
    Male | 16 | 6 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 0 | 5
  United States | 26 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Efficacy in Young Children Implanted Bilaterally With MED-EL COMBI 40+ / PULSARCI100/SONATATI100 Cochlear Implant Systems
Description: Speech perception scores will be compared pre-operatively and postoperatively.
Time Frame: 60 months post initial stimulation
Population: Pre- and post-operative data were not collected for this outcome measure and thus no data is reported here
Arm/Group | Bilateral | Unilateral
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Language Acquisition Over Time in Bilaterally Implanted Children.
Description: Scores over time on the MacArthur communicative development inventory.
Time Frame: 60 months post initial activation
Population: Pre- and post-operative data were not collected for this outcome measure and thus no data is reported here
Arm/Group | Bilateral | Unilateral
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Speech Production Over Time in Children Implanted Bilaterally With a MED-EL Cochlear Implant.
Description: Speech production scores over time on the Goldman-Fristoe test of articulation and the Kaufman speech praxis test for children.
Time Frame: 5 years
Population: Pre- and post-operative data were not collected for this outcome measure and thus no data is reported here.
Arm/Group | Bilateral | Unilateral
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through the study endpoint ( 5 years postoperatively) for each subject. However, due to early termination of the study the endpoint was not reached, and participants were followed for an average of 3 years postoperatively.
Description: Definitions do not differ
Arm/Group | Bilateral | Unilateral
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/31 | 0/6
Other Adverse Events (participants affected / at risk) | 4/31 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral (N=31) | Unilateral (N=6)
high fever during surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Surgery aborted due to high fever.
Device failure due to impact (Ear and labyrinth disorders) | 1 (1) | 0 (0) — head trauma which led to device failure
Device failure (Ear and labyrinth disorders) | 4 (4) | 0 (0) — Electrode failure determined by device telemetry and/or intermittent responsiveness
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral (N=31) | Unilateral (N=6)
Changes in device telemetry (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Protocol was terminated due to inability to find unilateral matches.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less